CLINICAL TRIAL: NCT06210737
Title: A Study to Evaluate Persistence of Immunity of PCV13 in Healthy Population Aged 2 Months，7 Months-5 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Minhai Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014L00987-1
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 months group (Other)
  Interventions: Biological: PCV13
- 7-11 months group (Other)
  Interventions: Biological: PCV13
- 12-23 months group (Other)
  Interventions: Biological: PCV13
- 2-5 years old group (Other)
  Interventions: Biological: PCV13

INTERVENTIONS:
Biological: PCV13 — 3 doses of PCV13 intramuscularly at Months 0, 2, and 4 and a booster dose at Month 10
  Arms: 2 months group
Biological: PCV13 — 2 doses of PCV13, and a booster dose
  Arms: 7-11 months group
Biological: PCV13 — 2 doses of PCV13
  Arms: 12-23 months group
Biological: PCV13 — single dose of PCV13
  Arms: 2-5 years old group

SUMMARY:
The goal of this clinical trial is to learn about persistence of immunity of PCV13 in healthy population aged 2 months, 7 months-5 years. The main questions it aims to answer are the percentage of subjects reached the IgG level of ≥0.35 µg/mL, GMCs level for IgG antibody, and SAEs from one month to 12 months after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Those who have participated in the Phase III clinical study of Beijing Minhai PCV13 and have been fully vaccinated with Minhai PCV13;
* An informed consent was required to sign by their legal guardians;
* Volunteers and their legal guardians/caregivers were able to attend the study visit as required by the protocol.

Exclusion Criteria:

* Those who had any administration history of pneumococcal polysaccharide or conjugate vaccine after participating in the Phase III clinical study;
* Prior to enrollment, patients who had a history of pneumococcal infection with one or more of the well-defined PCV13 serotypes;
* The researchers shall judge the other conditions which might be not in compliance with the requirements of this clinical trial.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 621 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2022-11-13 (Actual)

PRIMARY OUTCOMES:
percentage of subjects reached the IgG level of ≥0.35 µg/mL | 2-5 years after the first dose
  evaluation time: two years after the first dose for 2-5 years old group, two and three years after the first dose for 12-23 months group, two, three and four years after the first dose for 7-11 months group, two, three, four and five years after the first dose for 2 months group.
GMCs level for IgG antibody | 2-5 years after the first dose
  evaluation time: two years after the first dose for 2-5 years old group, two and three years after the first dose for 12-23 months group, two, three and four years after the first dose for 7-11 months group, two, three, four and five years after the first dose for 2 months group.
Serious Adverse Events (SAE) | one months to 12 months after the last injection

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Li G, Ren T, Zhang H, Ti J, Chang X, Yin S, Guan Y, Liu G, Liang Q, Liu J. Persistence of immunity in children aged 2 months and 7 months - 5 years old after primary immunization with 13-valent pneumococcal conjugate vaccine. Vaccine. 2024 Oct 24;42(24):126209. doi: 10.1016/j.vaccine.2024.126209. Epub 2024 Aug 31. PMID 39217777